CLINICAL TRIAL: NCT00408148
Title: A Randomized, Double-blind, Two Arm, Parallel, Placebo Controlled Study of Rimonabant 20 mg Effect on High Density Lipoprotein Kinetics in Patients With Abdominal Obesity and Additional Cardiometabolic Risk Factors
Brief Title: High Density Lipoprotein Turnover
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision has been taken in light of recent demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIMON_C_01346; EUDRACT # : 2006-001716-71
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 2 (Placebo Comparator): Administration of one rimonabant placebo tablet once daily in the morning
  Interventions: Drug: Placebo
- 1 (Experimental): Administration of one tablet containing 20 mg of active rimonabant once daily in the morning
  Interventions: Drug: Rimonabant

INTERVENTIONS:
Drug: Placebo — Undistinguishable placebo tablets
  Arms: 2
Drug: Rimonabant — White film-coated, for oral administration containing 20 mg of active rimonabant
  Arms: 1

SUMMARY:
The objective of the study is to evaluate the effect of Rimonabant 20mg in comparison to placebo, on HDL and VLDL lipoprotein kinetics, over a 12 months period.

Primary objectives:

* To assess effect of Rimonabant on HDL ApoA-I fractional catabolic rate (FCR).

Secondary objectives:

* To assess effect of Rimonabant on HDL ApoA-I production rate (PR) and on other lipoprotein kinetics.
* To assess effect of Rimonabant on lipids, glycemic and inflammatory parameters
* To assess effect of Rimonabant on body composition
* To assess safety of Rimonabant

ELIGIBILITY:
Inclusion Criteria:

* Abdominally obese patients with additional cardiometabolic risk factors
* Females must be post-menopausal
* BMI > 27 kg/m² and < 40 kg/m²
* Men or women with abdominal obesity according to NCEP/ATPIII criteria: Waist Circumference > 88 cm in women; > 102 cm in men
* With at least one lipid abnormality defined as:
* Fasting Triglycerides level > 1.7 mmol/L (150 mg/dL) and < 4.5 mmol/L (400 mg/dL)
* HDL < 1.03 mmol/L (40 mg/dL) in men and < 1.29 mmol/L (50 mg/dL) in women

Exclusion Criteria:

* HDL ≤ 0.60 mmol/L (23 mg/dl)
* Plasma LDL-Cholesterol > 155 mg/dl (4.00 mmol/L) or total cholesterol 250 mg/dl (> 6.5mmol/L) or genetic hyperlipidaemia
* Fasting triglycerides > 400 mg/dL (4.5 mmol/L)
* Known heterozygous or homozygous familial hypercholesterolaemia or know type III hyperlipoproteinaemia (familial dysbetalipoproteinaemia)
* ApoE2/E2 homozygosity, Apo E4/E4 homozygosity
* Type 2 diabetes treated with oral agents and/or insulin
* Diet treated type 2 diabetic patients with HbA1c ≥ 7%
* History of cardio vascular disease
* Systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 95 mmHg.
* Very low-calorie diet (1200 calories a day or less) or history of surgical procedures for weight loss (e.g., stomach stapling, bypass)
* Body weight fluctuation > 5 Kg during the previous 3 months
* History of bulimia or anorexia nervosa by DSM-IV criteria
* Presence of any clinically significant endocrine disease according to the investigator, Cushing syndrome, obesity secondary to hypothalamic/pituitary disorder.
* Abnormal TSH and free T4 at baseline (Patients treated with thyroid replacement therapy must be on fixed and stable dose for at least 3 months prior to screening and must be in euthyroïd status.)
* Severe hepatic impairment known by the investigator or AST or ALT > 3 times the ULN at screening.
* Known severe renal dysfunction (creatinine clearance < 30 ml/min) or urine analysis (performed at screening by dipstick) showing 2+ or more protein
* Presence of any condition (medical, including clinically significant abnormal laboratory test, psychological, social or geographical) actual or anticipated that the investigator feels would compromise the patient safety or limit his/her successful participation to the study
* Patient treated for epilepsy
* Ongoing major depressive illness
* Uncontrolled psychiatric illness
* History of alcohol and/or drug abuse
* Smoker or smoking cessation within the past 3 months
* Marijuana or hashish users
* Previous participation in a Rimonabant study or to any other clinical trial within 4 weeks to study start
* Hypersensitivity/intolerance to the active substance or to any of the excipients such as lactose
* Blood donation within the past 3 months prior to the study or planned during the study or within the 3 months from the study completing
* Recent history of active peptic ulcer
* Willebrand disease or other hemorrhagic diatheses
* Administration of any of the following within 3 months prior to screening visit and susceptible to be prescribed during the study treatment period:
* Lipid-lowering drugs intake
* Anti obesity drugs
* Other drugs for weight reduction (phentermine, amphetamines)
* Herbal preparations for weight reduction
* Other drugs known to affect lipid metabolism: retinoids, antiretroviral, estrogens and hormone replacement therapy, cyclosporine, glitazones, benfluorex, fish oils, plant sterols.
* Thiazids (including fixed combination) at daily dose higher than 12.5 mg
* Unselective beta-blockers
* Prolonged use (more than one week) of systemic corticosteroids, neuroleptics
* Anticoagulants
* Ongoing antidepressive treatment

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The fractional catabolic rate (FCR) of HDL ApoA-I | After 12 months of treatment.

SECONDARY OUTCOMES:
Production Rate (PR) of HDL ApoA-I and A-II, (FCR) of HDL ApoA-II | All across the study
PR and FCR of VLDL1 and VLDL2 Apo B, VLDL1 and VLDL2 TG, IDL Apo B and LDL Apo B | All across the study
Variation in ApoA-I, ApoA-II, Lp-AI, Lp-AII, pre-beta-HDL HDL2a, HDL2b, HDL3a, HDL3b, HDL3c, Apo B, Apo C III, TG, LDL-C, HDL-C levels | All across the study
Variation in Glucose, insulin, HbA1c, leptin, adiponectin | All across the study
Variation in hs-CRP, TNF-alpha, CETP, PLTP and LCAT activities, lipoprotein and hepatic lipase activities in post-heparin plasma | All across the study
Variation in whole body fat | All across the study
Variation in abdominal sub-cutaneous and visceral fat | All across the study
Variation in liver fat | All across the study
Variation in blood pressure | All across the study
Variation in body weight, waist circumference, waist/hip ratio | From the beginning to the end of the study
CE/TG ratio in HDL | All across the study
Adverse events | From the beginning to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Pilorget, Study Director — Sanofi
Locations (4):
- Sanofi-Aventis Administrative Office, North Ryde, Australia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Guildford, United Kingdom

REFERENCES:
- [Derived] Verges B, Adiels M, Boren J, Barrett PH, Watts GF, Chan D, Duvillard L, Soderlund S, Matikainen N, Kahri J, Robin I, Taskinen MR. Interrelationships between the kinetics of VLDL subspecies and HDL catabolism in abdominal obesity: a multicenter tracer kinetic study. J Clin Endocrinol Metab. 2014 Nov;99(11):4281-90. doi: 10.1210/jc.2014-2365. Epub 2014 Jul 31. PMID 25077901